CLINICAL TRIAL: NCT02077582
Title: Longitudinal Observation of Brain Ischemia and Blood Brain Barrier Permeability in the Acute Phase of Ischemic Stroke
Brief Title: Longitudinal MRI Examinations of Patients With Brain Ischemia and Blood Brain Barrier Permeability
Acronym: LOBI-BBB
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Charite University, Berlin, Germany (Other)
Collaborators: German Federal Ministry of Education and Research (Other Government)
Responsible Party: Principal Investigator, Jochen B. Fiebach, MD, Charite University, Berlin, Germany
Other Study IDs: LOBI-BBB; EA1/200/13 (Other: Ethics Comittee of the Charité Universitätsmedizin Berlin)
Record Dates: First submitted 2014-02-23; First posted 2014-03-04 (Estimated); Last update posted 2014-03-04 (Estimated); Status verified 2014-03

CONDITIONS: Cerebral Stroke
Keywords: acute ischemic stroke
MeSH Terms: conditions — Stroke; Ischemic Stroke

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — 2x 2ml plasma and 2x 2ml serum per patient
Oversight: Data Monitoring Committee: No

SUMMARY:
The objective of this trial is to visualize blood brain barrier function and metabolic changes in the first days after ischemic stroke with new investigational MRI sequences.

DETAILED DESCRIPTION:
In this study the investigators will be examining acute ischemic stroke patients on the first and second day after symptom onset using repetitive MRI examinations to visualize blood brain barrier function and metabolic changes of the brain in 5 sub-projects, each containing a specific MRI protocol with one of the following new MRI sequences:

1. T1-Dynamics (measuring disruptions of the blood-brain barrier)
2. pH-imaging (measuring metabolic changes, acidosis)
3. Resting-state MRI (measuring changes in the cerebral perfusion)
4. Quantitative MRI-Angiography (quantification of blood flow in single vessels)
5. Diffusion Tensor Imaging (DTI) for patients with Anterior Choroidal Artery (AChA)-Infarcts (quantification of damage of white matter tracts)

Each sub-projects will be conducted in blocks of a specific time span. Morphological outcome will be assessed at day 5-7. Clinical outcome will be assessed at day 5-7 and day 90. The association of the new imaging parameter with the clinical and morphological outcome measures will be analysed. No specific intervention is assigned to the subjects by the investigators of the study.

ELIGIBILITY:
Inclusion Criteria:

* Suspected stroke or transient ischemic attack (TIA) within 24h from symptom onset

Exclusion Criteria:

* MRI contraindication, age < 18 years, intracranial hemorrhages

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Primary care clinic. Patients presenting with acute (<24h) transient ischemic attack or stroke at the emergency ward, Charité Campus Benjamin Franklin
Sampling Method: Non-Probability Sample
Enrollment: 410 (Estimated)
Dates: Start 2013-09; Primary Completion 2018-09 (Estimated); Study Completion 2018-12 (Estimated)

PRIMARY OUTCOMES:
clinical outcome measured with the National Institutes of Health Stroke Scale (NIHSS) | on follow-up examination day 5-7
clinical outcome measured with the modified Rankin Scale (mRS) | on day 90
  conducted as telephone interview

SECONDARY OUTCOMES:
final lesion volume (measured on FLAIR images) | on follow-up examination day 5-7

OTHER OUTCOMES:
volumes of hypoperfusion on resting state-MRI perfusion maps | on follow-up examinations day 1 and 2
  outcome measure for resting state-MRI sub-project only
blood flow parameters in occluded, contralateral and (partially) recanalized vessels | on follow-up examinations day 1 and 2
  outcome measure for quantitative Angiography sub-project only
pH values in the region of diffusion restriction and in the region of final infarct | on follow-up examinations day 1 and 2
  outcome measure for the pH-Imaging sub-project only
quantified values for contrast agent enhancement in the stroke lesion and on the contralateral side | on follow-up examination day 1 and 2
  outcome measure for the T1-Dynamic sub-project only

CONTACTS AND LOCATIONS:
Locations (1):
- Center for Stroke Research Berlin, Charité Universitätsmedizin Berlin, Campus Benjamin Franklin, Berlin, State of Berlin, Germany

REFERENCES:
- [Derived] Fan AP, Khalil AA, Fiebach JB, Zaharchuk G, Villringer A, Villringer K, Gauthier CJ. Elevated brain oxygen extraction fraction measured by MRI susceptibility relates to perfusion status in acute ischemic stroke. J Cereb Blood Flow Metab. 2020 Mar;40(3):539-551. doi: 10.1177/0271678X19827944. Epub 2019 Feb 7. PMID 30732551
- [Derived] Villringer K, Florczak-Rzepka M, Grittner U, Brunecker P, Tepe H, Nolte CH, Fiebach JB. Characteristics associated with outcome in patients with first-ever posterior fossa stroke. Eur J Neurol. 2018 Jun;25(6):818-824. doi: 10.1111/ene.13596. Epub 2018 Mar 25. PMID 29431878
- [Derived] Ganeshan R, Nave AH, Scheitz JF, Schindlbeck KA, Haeusler KG, Nolte CH, Villringer K, Fiebach JB. Assessment of thrombus length in acute ischemic stroke by post-contrast magnetic resonance angiography. J Neurointerv Surg. 2018 Aug;10(8):756-760. doi: 10.1136/neurintsurg-2017-013454. Epub 2017 Nov 18. PMID 29151041
- [Derived] Khalil AA, Ostwaldt AC, Nierhaus T, Ganeshan R, Audebert HJ, Villringer K, Villringer A, Fiebach JB. Relationship Between Changes in the Temporal Dynamics of the Blood-Oxygen-Level-Dependent Signal and Hypoperfusion in Acute Ischemic Stroke. Stroke. 2017 Apr;48(4):925-931. doi: 10.1161/STROKEAHA.116.015566. Epub 2017 Mar 8. PMID 28275197
- [Derived] Villringer K, Sanz Cuesta BE, Ostwaldt AC, Grittner U, Brunecker P, Khalil AA, Schindler K, Eisenblatter O, Audebert H, Fiebach JB. DCE-MRI blood-brain barrier assessment in acute ischemic stroke. Neurology. 2017 Jan 31;88(5):433-440. doi: 10.1212/WNL.0000000000003566. Epub 2016 Dec 28. PMID 28031392